CLINICAL TRIAL: NCT00002879
Title: A PHASE II TRIAL OF 2-CDA IN PREVIOUSLY TREATED OR UNTREATED PATIENTS WITH MANTLE CELL LYMPHOMA (MCL)
Brief Title: Cladribine in Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-958053; NCI-2012-02249 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000065179 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: mantle cell lymphoma; stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cladribine (Experimental): Patients receive cladribine (2-chlorodeoxyadenosine; 2-CdA) daily for 5 days every 4 weeks for a maximum of 6 courses; response is assessed after every 2 courses. Patients in complete remission or with stable disease discontinue treatment and are followed; those with disease progression at any time are removed from study. Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and annually for 2 years.
  Interventions: Drug: cladribine

INTERVENTIONS:
Drug: cladribine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effects of cladribine in previously treated or untreated patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of cladribine (2-chlorodeoxyadenosine; 2-CdA) as treatment for mantle cell lymphoma (MCL) either as initial therapy or for relapsed/refractory disease. II. Determine by flow cytometry immunophenotyping of blood lymphocytes the number of patients with peripheral blood involvement at the time of diagnosis and compare the presence or absence of peripheral blood involvement with response data. III. Detect rearrangements involving the bcl-1 gene and immunoglobulin heavy chain locus by molecular techniques (e.g., polymerase chain reaction, Southern blotting, or in situ hybridization), and compare these results with immunohistochemical demonstration of bcl-1 protein expression. VI. Determine the proliferative rate of MCL by immunohistochemistry and DNA content flow cytometry. V. Summarize the toxic effects associated with this treatment.

OUTLINE: Patients receive cladribine (2-chlorodeoxyadenosine; 2-CdA) daily for 5 days every 4 weeks for a maximum of 6 courses; response is assessed after every 2 courses. Patients in complete remission or with stable disease discontinue treatment and are followed; those with disease progression at any time are removed from study. Patients are followed every 2 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed mantle cell lymphoma (MCL) requiring therapy NCCTG pathology review required - Repeat biopsy is required for previously treated patients with previously biopsy proven MCL who relapse after achieving a partial or complete remission - Rebiopsy is not required for patients with: Progression of previously biopsy proven MCL who have not received therapy since the diagnostic biopsy OR Previously biopsy proven MCL who progress or achieve less than a partial remission following initial therapy Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST no greater than 3 times normal (5 times normal with liver involvement) Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No uncontrolled hypertension No unstable angina No active congestive heart failure No myocardial infarction within 6 months No serious uncontrolled arrhythmia Other: No active or uncontrolled infection No HIV antibody No medical or psychiatric condition that precludes participation No malignancy in the past 5 years, except carcinoma in situ of the cervix, resected basal cell or squamous cell carcinomas of the skin, or prostate cancer that is in remission following a radical retropubic prostatectomy or radiation therapy No pregnant or nursing women Negative pregnancy test required of fertile women within 7 days prior to entry Effective contraception required of fertile patients throughout study and at least 30 days thereafter

PRIOR CONCURRENT THERAPY: Recovered from any reversible acute toxic effects of previous therapy Biologic therapy: Not specified Chemotherapy: At least 4 weeks since chemotherapy (8 weeks since nitrosoureas or mitomycin) No prior fludarabine, pentostatin, or cladribine Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to greater than 25% of bone marrow Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1996-11; Primary Completion 2005-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Overall response | Up to 4 years
Overall survival | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: David J. Inwards, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (20):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Inwards DJ, Fishkin PA, Hillman DW, Brown DW, Ansell SM, Kurtin PJ, Fonseca R, Morton RF, Veeder MH, Witzig TE. Long-term results of the treatment of patients with mantle cell lymphoma with cladribine (2-CDA) alone (95-80-53) or 2-CDA and rituximab (N0189) in the North Central Cancer Treatment Group. Cancer. 2008 Jul 1;113(1):108-16. doi: 10.1002/cncr.23537. PMID 18470909
- [Result] Inwards D, Brown D, Fonseca R, et al.: NCCTG Phase II trial of 2-chlorodeoxyadenosine (2-CDA) as initial therapy for mantle cell lymphoma. A well-tolerated treatment with promising activity. Blood 94(10 suppl 1): A-2930, 660a, 1999.